CLINICAL TRIAL: NCT03304457
Title: Effect of Lurasidone Vs Olanzapine on Neurotrophic Biomarkers and Cardiometabolic Parameters in First Episode Untreated Schizophrenia: A Randomized, Open Label, Active Controlled Study
Brief Title: Lurasidone Vs Olanzapine on Neurotrophic Biomarkers and Cardiometabolic Parameters in Unmedicated Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Dr. Monalisa Jena, M.D., Assistant Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T/IM-F/17-18/29
Record Dates: First submitted 2017-10-03; First posted 2017-10-09 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Schizophrenia
Keywords: Lurasidone; Olanzapine; Brain derived neurotrophic factor; Nerve growth factor; Neurotrophin 3
MeSH Terms: conditions — Schizophrenia; Hereditary Sensory and Autonomic Neuropathies | interventions — Olanzapine; Lurasidone Hydrochloride

STUDY DESIGN:
Intervention Model Description: A randomized, open label, active controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olanzapine (Active Comparator): Olanzapine will be prescribed at a dose of 10mg once daily orally for 6 weeks
  Interventions: Drug: Olanzapine
- Lurasidone (Experimental): Lurasidone will be prescribed at a dose of 80mg/day once daily orally for 6 weeks
  Interventions: Drug: Lurasidone

INTERVENTIONS:
Drug: Olanzapine — Olanzapine 10mg once daily orally for 6 weeks
  Arms: Olanzapine
Drug: Lurasidone — Lurasidone 80mg once daily orally for 6 weeks
  Arms: Lurasidone

SUMMARY:
Schizophrenia (SCZ) is a chronic, severe and disabling mental disorder with unclear etiology and pathophysiology concerned with neuro-developmental,neurodegenerative abnormalities and cognitive impairmentslinked to behavioural changes.According to neurotrophic hypothesis, the changes result due to the abnormal regulation of neurotrophic factor, especially the decreased serum brain derived neurotrophic factor (BDNF) validated by several meta-analyses. However, the regulation of nerve growth factor (NGF) in SCZ remains unclear because of the inconsistent findings from the previous clinical studies.

Lurasidone is a novel antipsychotic drug approved for adult SCZ and for affective symptomatology & cognitive deficits. Principal advantages over some other second-generation antipsychotics are its highly favourable metabolic profile and once daily dosing regimen. Some of the studies indicate that risperidone, olanzapine, clozapine & aripiprazole might not alter BDNF levels, at least within 8 weeks of treatment.While other two studies with olanzapine suggest that BDNF might influence the response to monotherapy in SCZ patients.All these previous studies are non-conclusive & contradictory to each other which draw our attention for doing the research further to reach a conclusive result about the effect of olanzapine and lurasidone on neurotrophic biomarkers in SCZ.

DETAILED DESCRIPTION:
Schizophrenia (SCZ) is a chronic, severe and disabling mental disorder with unclear aetiology and pathophysiology concerned with neuro-developmental,neurodegenerative abnormalities and cognitive impairments linked to behavioural changes.According to neurotrophic hypothesis, the changes result due to the abnormal regulation of neurotrophic factor, especially the decreased serum brain derived neurotrophic factor (BDNF) validated by several meta-analyses. However, the regulation of nerve growth factor (NGF) in SCZ remains unclear because of the inconsistent findings from the previous clinical studies.

Lurasidone is a novel antipsychotic drug approved for adult SCZ and for affective symptomatology & cognitive deficits. Principal advantages over some other second-generation antipsychotics are its highly favourable metabolic profile and once daily dosing regimen. Some of the studies indicate that risperidone, olanzapine, clozapine & aripiprazole might not alter BDNF levels, at least within 8 weeks of treatment.While other two studies with olanzapine suggest that BDNF might influence the response to monotherapy in SCZ patients.All these previous studies are non-conclusive & contradictory to each other which draw our attention for doing the research further to reach a conclusive result about the effect of olanzapine and lurasidone on neurotrophic biomarkers in SCZ.

Most of the antipsychotic drugs prescribed for SCZ are based on the dopamine hypothesis. In recent times, neurotrophic hypothesis gained importance in the pathophysiology of SCZ. So, our study may enable psychiatrist to choose a better antipsychotic drug having effect on both dopamine as well as neurotrophic factors. Previously there were no studies on effect of lurasidone on neurotrophic factors in SCZ & also there was no head-on comparison of lurasidone and olanzapine

ELIGIBILITY:
Inclusion Criteria:

* All treatment naive patients clinically diagnosed first episode of SCZ according to ICD-10
* Patients of either sex with age range 18-45 years
* Treatment naïve patients

Exclusion Criteria:

* Other Psychotic spectrum disorders (F21- F29)
* Highly agitated/ violent/ suicidal patients who need immediate treatment
* Patients with comorbid substance abuse except Nicotine use or history of organicity
* Patients with known history of diabetes mellitus, hypertension or any long standing significant medical illness/ significant neurological impairment/ clinical observable mental retardation
* Pregnant and nursing women

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-25 (Actual)

PRIMARY OUTCOMES:
Serum brain derived neurotrophic factor (BDNF) | 6 weeks
  the change in serum level of BDNF from baseline after treatment with lurasidone or olanzapine

SECONDARY OUTCOMES:
serum nerve growth factor (NGF) | 6 weeks
  the change in serum level of NGF from baseline after treatment with lurasidone or olanzapine
Serum Neurotrophin 3 (NT3) | 6 weeks
  the change in serum level of NT3 from baseline after treatment with lurasidone or olanzapine
PANSS score | 6 weeks
  To determine the association (if any) between change in serum neurotrophic factor and PANSS score
Social and occupational functioning assessment scale (SOFAS) | 6 weeks
  To determine the association (if any) between change in serum neurotrophic factor and SOFAS (Social and occupational functioning assessment scale) score
Serum hsCRP | 6 weeks
  to assess cardiovascular risk in schizophrenia
Serum Insulin | 6 weeks
  to assess insulin resistance
LDL/HDL ratio | 6 weeks
  to assess dyslipidemia and cardiovascular risk
Fasting blood sugar | 6 weeks
  to assess dysglycemia
Glycosylated Hemoglobin (HbA1c) | 6 weeks
  to assess dysglycemia
High Density Lipoprotein (HDL) | 6 week
  to assess dyslipidemia
Low Density Lipoprotein (LDL) | 6 week
  to assess dyslipidemia
Very Low Density Lipoprotein (VLDL) | 6 week
  to assess dyslipidemia
Serum Triglyceride | 6 weeks
  to assess dyslipidemia

CONTACTS AND LOCATIONS:
Overall Officials: Debasish Hota, MD, DM, Study Director — Professor & Head
Locations (1):
- AIIMS, Bhubaneshwar, Odisha, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van Os J, Rutten BP, Poulton R. Gene-environment interactions in schizophrenia: review of epidemiological findings and future directions. Schizophr Bull. 2008 Nov;34(6):1066-82. doi: 10.1093/schbul/sbn117. Epub 2008 Sep 12. PMID 18791076
- [Result] Gejman PV, Sanders AR, Kendler KS. Genetics of schizophrenia: new findings and challenges. Annu Rev Genomics Hum Genet. 2011;12:121-44. doi: 10.1146/annurev-genom-082410-101459. PMID 21639796
- [Result] Owen MJ, O'Donovan MC, Thapar A, Craddock N. Neurodevelopmental hypothesis of schizophrenia. Br J Psychiatry. 2011 Mar;198(3):173-5. doi: 10.1192/bjp.bp.110.084384. PMID 21357874
- [Result] Ashe PC, Berry MD, Boulton AA. Schizophrenia, a neurodegenerative disorder with neurodevelopmental antecedents. Prog Neuropsychopharmacol Biol Psychiatry. 2001 May;25(4):691-707. doi: 10.1016/s0278-5846(01)00159-2. PMID 11383973
- [Result] Perez-Neri I, Ramirez-Bermudez J, Montes S, Rios C. Possible mechanisms of neurodegeneration in schizophrenia. Neurochem Res. 2006 Oct;31(10):1279-94. doi: 10.1007/s11064-006-9162-3. Epub 2006 Sep 28. PMID 17006758
- [Result] Matza LS, Buchanan R, Purdon S, Brewster-Jordan J, Zhao Y, Revicki DA. Measuring changes in functional status among patients with schizophrenia: the link with cognitive impairment. Schizophr Bull. 2006 Oct;32(4):666-78. doi: 10.1093/schbul/sbl004. Epub 2006 Jul 7. PMID 16829550
- [Result] Ahmed AO, Mantini AM, Fridberg DJ, Buckley PF. Brain-derived neurotrophic factor (BDNF) and neurocognitive deficits in people with schizophrenia: a meta-analysis. Psychiatry Res. 2015 Mar 30;226(1):1-13. doi: 10.1016/j.psychres.2014.12.069. Epub 2015 Jan 28. PMID 25681004
- [Result] Yoshimura R, Ueda N, Hori H, Ikenouchi-Sugita A, Umene-Nakano W, Nakamura J. Different patterns of longitudinal changes in plasma levels of catecholamine metabolites and brain-derived neurotrophic factor after administration of atypical antipsychotics in first episode untreated schizophrenic patients. World J Biol Psychiatry. 2010 Mar;11(2 Pt 2):256-61. doi: 10.3109/15622970802309617. PMID 20218790
- [Result] Yoshimura R, Hori H, Sugita A, Ueda N, Kakihara S, Umene W, Nakano Y, Shinkai K, Mitoma M, Ohta M, Shinkai T, Nakamura J. Treatment with risperidone for 4 weeks increased plasma 3-methoxy-4-hydroxypnenylglycol (MHPG) levels, but did not alter plasma brain-derived neurotrophic factor (BDNF) levels in schizophrenic patients. Prog Neuropsychopharmacol Biol Psychiatry. 2007 Jun 30;31(5):1072-7. doi: 10.1016/j.pnpbp.2007.03.010. Epub 2007 Mar 24. PMID 17459549
- [Result] Hori H, Yoshimura R, Yamada Y, Ikenouchi A, Mitoma M, Ida Y, Nakamura J. Effects of olanzapine on plasma levels of catecholamine metabolites, cytokines, and brain-derived neurotrophic factor in schizophrenic patients. Int Clin Psychopharmacol. 2007 Jan;22(1):21-7. doi: 10.1097/YIC.0b013e3280103593. PMID 17159456
- [Result] Nikolac Perkovic M, Nedic Erjavec G, Zivkovic M, Sagud M, Uzun S, Mihaljevic-Peles A, Kozumplik O, Muck-Seler D, Pivac N. Association between the brain-derived neurotrophic factor Val66Met polymorphism and therapeutic response to olanzapine in schizophrenia patients. Psychopharmacology (Berl). 2014 Sep;231(18):3757-64. doi: 10.1007/s00213-014-3515-4. Epub 2014 Mar 5. PMID 24595507
- [Result] Gonzalez-Pinto A, Mosquera F, Palomino A, Alberich S, Gutierrez A, Haidar K, Vega P, Barbeito S, Ortiz A, Matute C. Increase in brain-derived neurotrophic factor in first episode psychotic patients after treatment with atypical antipsychotics. Int Clin Psychopharmacol. 2010 Jul;25(4):241-5. doi: 10.1097/yic.0b013e328338bc5a. PMID 20568658
- [Derived] Jena M, Mishra A, Mishra BR, Nath S, Maiti R. Effect of lurasidone versus olanzapine on cardiometabolic parameters in unmedicated patients with schizophrenia: a randomized controlled trial. Psychopharmacology (Berl). 2020 Nov;237(11):3471-3480. doi: 10.1007/s00213-020-05628-3. Epub 2020 Aug 1. PMID 32740676
- [Derived] Jena M, Ranjan R, Mishra BR, Mishra A, Nath S, Sahu P, Meher BR, Srinivasan A, Maiti R. Effect of lurasidone vs olanzapine on neurotrophic biomarkers in unmedicated schizophrenia: A randomized controlled trial. J Psychiatr Res. 2019 May;112:1-6. doi: 10.1016/j.jpsychires.2019.02.007. Epub 2019 Feb 12. PMID 30782512